CLINICAL TRIAL: NCT00424619
Title: A Randomised, Controlled Comparison of Vitamin D Strategies is Acute Hip Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Dr. Alexandra Papaioannou, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-449; P1975
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2012-05

CONDITIONS: Hip Fracture
Keywords: Vitamin D; Hip fracture; Optimal level; Deficiency; Functional muscle strength
MeSH Terms: conditions — Hip Fractures | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 50 000 IU Vitamin D2
  Interventions: Drug: Vitamin D2
- 2 (Active Comparator): 100 000 IU Vitamin D2
  Interventions: Drug: Vitamin D2
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D2 — 50 000 IU vitamin D2, one time bolus dose
  Other Names: Ostoforte
  Arms: 1
Drug: Vitamin D2 — 100 000 IU vitamin D2, one time bolus dose
  Other Names: Ostoforte
  Arms: 2
Drug: Placebo — Placebo, 1 time bolus dose
  Arms: 3

SUMMARY:
The purpose of the study is to determine the best dose of Vitamin D to give to hip fracture patients to achieve the optimal therapeutic level.

DETAILED DESCRIPTION:
Low Vitamin D levels can cause faster bone loss and increase the risk of having a fracture. Patients who experience a hip fracture have low levels of Vitamin D. It is not clear how much Vitamin D must be taken in order to reach this optimal level.

Serum 25-hydroxyvitamin D3 (25-OHD) concentrations are the recognized functional status indicator for vitamin D. Although there is no clear consensus, vitamin D 'insufficiency' has been considered in the range of 25- 75/80 nmol/L. Patients with acute hip fracture are at high risk for a recurrent hip fracture or other fragility fractures (and falls) and are a group who should be targeted for osteoporosis treatment (i.e. Bisphosphonate or other antiresorptive). Before fracture patients start on a bisphosphonate, however, an important consideration is whether 25-OHD levels are at a therapeutic level (>75 nmol/l and less than 150-200 nmol/L). Case-control studies indicate that older people who experience a hip fracture have lower serum concentrations of 25-OHD than do those without a fracture. In cross-sectional studies, the majority of patients with hip fracture are considered to have insufficient vitamin D levels. Although the benefits of supplementing patients with at least 800 to 1000 IU/day Vitamin D3 may be recognized, there is little information available to guide physicians regarding the appropriate management of hip fracture patients who may be severely Vitamin D deficient, particularly in acute hip fracture patients. Few studies have examined whether high dose vitamin D (i.e. 50,000 IU or greater/week) offers an advantage over smaller, routinely prescribed doses (i.e. 800 or 1000 IU), particularly in hip fracture patients.

The purpose of this study is to determine the number of hip fracture patients reaching an optimal level of vitamin D comparing between three different Vitamin D dose strategies:

A. 50,000 D2 oral bolus followed by 800 IU D3 daily B. 100,000 D2 oral bolus followed by 800 IU D3 daily C. 800 IU D3 daily

The Vitamin D strategies will be administered over 3-months in acute hip fracture patients. The proportion of patients reaching an optimal level of 25-OHD (>75 nmol/L) will be determined.

Secondary measures include the Timed Up and Go test, and 2 Minute Walk Test to compare the effects of the Vitamin D supplementation strategies on functional and muscle strength scales.

ELIGIBILITY:
Inclusion Criteria:

* Fragility hip fracture patient
* Previous Vitamin D supplementation is okay.

Exclusion Criteria:

* Patients with pathological fracture secondary to malignancy or intrinsic bone disease (eg. Paget's disease)
* Cancer in the past 10 years likely to metastasize to bone
* Renal insufficiency (creatinine <30 mls/min)
* Hypercalcemia (primary hyperparathyroidism; granulomatous diseases; drug-induced such as lithium, thiazides), hypocalcemia, hypercalciuria, fracture or stroke within the last 3 months
* Hormone replacement therapy, calcitonin, fluoride, or bisphosphonates during the previous 24 months
* Pre-existing bone abnormality
* Renal stones in past 10 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, M.D., M.Sc., Principal Investigator — McMaster University

REFERENCES:
- [Derived] Papaioannou A, Kennedy CC, Giangregorio L, Ioannidis G, Pritchard J, Hanley DA, Farrauto L, DeBeer J, Adachi JD. A randomized controlled trial of vitamin D dosing strategies after acute hip fracture: no advantage of loading doses over daily supplementation. BMC Musculoskelet Disord. 2011 Jun 20;12:135. doi: 10.1186/1471-2474-12-135. PMID 21689448

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 000 IU Vitamin D2: 50 000 IU Vitamin D2 at beginning of study and 1000IU vitamin D3 for 90 days
- 100 000 IU Vitamin D2: 100 000 IU Vitamin D2 at beginning of study and 1000IU vitamin D3 for 90 days
- Placebo: Placebo at beginning of study and 1000IU vitamin D3 for 90 days
Period: Baseline
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Started | 22 | 22 | 21 (n=21 but one participant was lost as a screen failure)
Completed | 22 | 22 | 20
Not Completed | 0 | 0 | 1
Period: 4 Week
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Started | 18 | 17 | 17
Completed | 18 | 17 | 17
Not Completed | 0 | 0 | 0
Period: 3 Month
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Started | 12 | 18 | 17
Completed | 12 | 18 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 20 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.9 (8.7) | 73.9 (12.4) | 78.5 (10.3) | 78.43 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 13 | 36
  Male | 7 | 14 | 7 | 28
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 22 | 20 | 64

OUTCOME MEASURES:

1. Secondary Outcome: Functional Assessment Using the Timed Up and Go (TUG) Test After 3 Months
Description: The Timed Up and Go (TUG) was collected for patients who attended the 3-month clinic appointment by study coordinators or for patients who attended the rehabilitation unit this is routinely collected and was abstracted from chart. The TUG was conducted using a standard armchair and a line marked 3-metres from the chair. Participants were given the following instructions (no physical assistance was given): "Rise from the chair, walk to the line on the floor, turn, return to the chair and sit down again". Scores are measured as time in seconds to complete the task.
Time Frame: 3 months
Population: The number of participants who completed the TUG test is lower than the number of participants who completed the primary outcome at this time point. Not everyone chose to complete the functional TUG test at this time point.
Measure: Mean (Full Range); unit: seconds
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 8 | 15 | 11
seconds | 26.2 [19.2 to 33.2] | 19.1 [14.1 to 24.1] | 18.1 [12.4 to 23.8]

2. Primary Outcome: 25-hydroxyvitamin D3 (25-OHD)
Description: Serum 25-hydroxyvitamin D3 (25-OHD) was measured at baseline, at discharge from hospital (approximately 4-weeks), and at a follow-up study visit at approximately 3-months.Baseline and 4-week blood samples were drawn in-hospital; venipunctures performed at 3-months were either in-hospital (if patient remained in acute care or rehabilitation) or at the out-patient clinic visit.Serum 25-OHD was analyzed with the DiaSorin, 25-hydroxyvitamin D radioimmunoassay (Stillwater, Minnesota 55082-0285, U.S.A) at the central laboratory with the exception of 3 patients (data analyzed at other laboratories).
Time Frame: Baseline, 4 weeks and 3 months
Population: Baseline data (n=59) was missing for two participants, and four outliers with 25-OHD taken at 6, 10 or 12 days were not included. 4-week data (n=50) was missing for 13 participants, and two outliers with 25-OHD taken at <13 days were not included. 3-month data (n=47) was missing for 18 participants.
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 20 | 21 | 18
nmol/L
  Baseline | 53.5 (34.8-58.6) [42.3 to 64.8] | 58.4 [47.3 to 69.5] | 46.7 [34.8 to 58.6]
  4-week | 84.5 [73.7 to 95.3] | 75.6 [64.5 to 86.8] | 69.3 [58.4 to 80.2]
  3-month | 84.2 [73.6 to 94.9] | 73.3 [64.5 to 82.1] | 86.7 [77.6 to 95.9]

3. Primary Outcome: Parathyroid Hormone (PTH)
Description: Baseline blood samples were drawn in-hospital. In additional PTH was accessed at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 22 | 22 | 20
pmol/L | 5.35 (3.01) | 5.10 (3.91) | 4.2 (2.12)

4. Primary Outcome: Calcium
Description: Baseline blood samples were drawn in-hospital. In additional Calcium was accessed at baseline and approximately 4 weeks.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 21 | 22 | 20
mmol/L
  Baseline | 2.10 (0.14) | 2.12 (0.11) | 2.08 (0.14)
  4 Weeks | 2.26 (0.17) | 2.31 (0.11) | 2.28 (0.15)

5. Primary Outcome: Phosphate
Description: Baseline blood samples were drawn in-hospital. In additional phosphate was accessed at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 22 | 22 | 20
mmol/L | 0.86 (0.22) | 0.97 (0.24) | 0.94 (0.27)

6. Primary Outcome: Alkaline Phosphatase
Description: Baseline blood samples were drawn in-hospital. In additional Alkaline Phosphatase was accessed at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 22 | 22 | 20
U/L | 98.6 (3.78) | 78.7 (26.2) | 79.4 (51.1)

7. Primary Outcome: Hemoglobin
Description: Baseline blood samples were drawn in-hospital. In additional hemoglobin was accessed at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 22 | 22 | 20
g/L | 102.2 (14.3) | 107.9 (17.4) | 108.6 (15.2)

8. Primary Outcome: Creatinine
Description: Baseline blood samples were drawn in-hospital. In additional creatinine was accessed at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 22 | 22 | 20
µmol/L | 70.5 (23.8) | 77.4 (26.1) | 73.7 (37)

9. Secondary Outcome: Functional Assessment Using the Two Minute Walk Test (2MWT)After 3 Months
Description: The 2MWT was collected for patients who attended the 3-month clinic appointment by study coordinators or for patients who attended rehabilitation, it was abstracted from their charts. The 2MWT test was given in a carpeted corridor and the subject was instructed to wear regular footwear and to use their customary walking aid. The distance the participant could comfortably walk in two-minutes (without physical assistance) was measured in metres.
Time Frame: 3 months
Population: The number of participants who completed the 2WT is lower than the number of participants who completed the primary outcome at this time point. Not everyone chose to complete the functional 2WT test at this time point.
Measure: Mean (Full Range); unit: meters
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Number analyzed (Participants) | 9 | 14 | 11
meters | 60.2 [41.2 to 79.1] | 80.3 [65.2 to 95.5] | 63.4 [45.4 to 81.5]

ADVERSE EVENTS:
Arm/Group | 50 000 IU Vitamin D2 | 100 000 IU Vitamin D2 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 3/22 | 1/20
Other Adverse Events (participants affected / at risk) | 2/22 | 0/22 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 000 IU Vitamin D2 (N=22) | 100 000 IU Vitamin D2 (N=22) | Placebo (N=20)
fractured hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edmea and Myocardial infarction (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
gangrenous left foot requiring amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 000 IU Vitamin D2 (N=22) | 100 000 IU Vitamin D2 (N=22) | Placebo (N=20)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Trip and fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distention, nausea, vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No